CLINICAL TRIAL: NCT06728696
Title: Peri-implant Tissue Changes Using Dual Zone Concept with Connective Tissue Graft Versus Concentrated Growth Factor (A Randomized Clinical Trial)
Brief Title: Peri-implant Tissue Changes Using Dual Zone Concept with Connective Tissue Graft Versus Concentrated Growth Factor
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1383
Record Dates: First submitted 2024-11-22; First posted 2024-12-11 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-09

CONDITIONS: Hopeless Tooth in Esthetic Zone; Loss of Soft and Hard Tissue Around Implant; Immediate Implant Placement
Keywords: Immediate implant; Esthetic zone; Connective Tissue Graft; Concentrated Growth Factor Graft

STUDY DESIGN:
Intervention Model Description: Randomized, parallel design, two arms clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to the type of the intervention and the whole-time frame of the study will be 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Test group): (Experimental): 17 patients with non-restorable tooth in the esthetic zone will receive atraumatic extraction followed by immediate implant placement with dual zone technique using concentrated growth factor graft.
  Interventions: Procedure: Immediate implant with with dual zone technique using concentrated growth factor graft.
- Group II (Control group): (Active Comparator): 17 patients with non-restorable tooth in the esthetic zone will receive atraumatic extraction followed by immediate implant placement with dual zone technique using connective tissue graft.
  Interventions: Procedure: Immediate implant with dual zone technique using connective tissue graft.

INTERVENTIONS:
Procedure: Immediate implant with with dual zone technique using concentrated growth factor graft. — In the test group, pouch technique + CGFG will be used. The CGFG will be packed in the split-thickness labial pouch between the labial bone plate and the overlying gingiva of the extraction socket. A convenient blood sample will be withdrawn from a peripheral venous blood from the patient using a specialized vacutaine. A standard, disposable, 10-ml non- anticoagulant tube and a matching centrifuge device was used. To prepare the CGFG, the centrifuge is accelerated for 30 seconds, then centrifuged at 2700 rpm for 2 minutes, 2400 rpm for 4 minutes, 2700 rpm for 4 minutes, and 3000 rpm for 3 minutes before being decelerated for 36 seconds to stop.
  Arms: Group I (Test group):
Procedure: Immediate implant with dual zone technique using connective tissue graft. — Patients assigned to the control group will receive pouch technique + CTG. Following implant placement, a split-thickness labial pouch between the labial bone plate and the overlying gingiva of the extraction socket will be performed using 15c mini blade to allow for the placement of a CTG. The pouch preparation will be extended apical beyond the muco-gingival junction and to the neighboring teeth mesiodistally. The CTG will be harvested from the palate with a thickness of 1.5 mm using single-incision technique, which was done approximately 2-3 mm apical to the gingival margin of the maxillary teeth and parallel to the palatal long axis. A resorbable suture will be used to first pierce the labial mucosa along with the periosteum at an apical part, which then exits from the sulcus. Afterward, the CTG will be tucked in the pouch, labial to the suture, and held at a coronal area by using the needle to pierce it from its inner surface toward the labial soft tissue. The knot will then be se
  Arms: Group II (Control group):

SUMMARY:
Tooth extraction not only alters the bony architecture of the alveolar ridge, but it also has an impact on the surrounding soft tissues. Post-extraction recovery of both hard and soft tissues occurs uneventfully, resulting in horizontal and vertical tissue loss, affecting prosthetic rehabilitation with dental implants or tooth-supported prosthesis.

Aim of the study:

The aim of this study is to evaluate volumetric soft tissue alterations as well as clinical, radiographic, and esthetic outcomes in dual zone technique (DZ) using CTG (Connective Tissue Graft) versus CGF (Concentrated Growth Factor) Graft following maxillary IIP (Immediate Implant Placement) in the esthetic zone.

Materials and methods:

20 patients with hopeless teeth requiring extraction in maxillary esthetic zone and requiring replacement with dental implants, will be enrolled and recruited from the outpatient clinic, faculty of dentistry, Ain Shams University according to the inclusion criteria. They will be randomly allocated into two equal groups. Group I (n=17) immediate implant placement with dual zone technique using concentrated growth factor graft and group II (n=17) immediate implant placement with dual zone technique using connective tissue graft. Pink esthetic score (PES) was measured 6 months after the final crown placement. At the respective times radiographic CBCT measurements, volumetric analysis, and clinical measurements will be taken. Postoperative medication will be prescribed to the patient and postoperative instructions will be explained in detail. Follow-up will be performed. Data collected will be tabulated and statistically analyzed.

DETAILED DESCRIPTION:
Maintaining the natural esthetic appearance, particularly in the esthetic zone, together with the volume and contour of the soft tissue in harmony with the surrounding teeth soft tissue, is believed to be critical. However, postponing implant placement until hard and soft tissues have fully healed usually necessitates additional surgical intervention steps, such as guided bone regeneration or ridge splitting, or implant placement in undesirable positions with a low esthetic appearance to overcome alveolar ridge resorption.

In clinical practice, immediate implant placement (IIP) in the esthetic zone has been regarded as an ongoing concern. Immediate implant placement (IIP) aims to minimize the duration of therapy overall, cost-effectiveness, and patient aesthetic expectations. However, the physician needs to be aware of potential risks and undesirable effects associated with this surgery, such as early implant loss and dimensional alterations in soft and hard tissues. Clinical research continues to advance to improve predictability and minimize the occurrence of undesirable consequences following IIP due to evolving patients' esthetic demands and expectations.

Over the years, numerous surgical techniques have been proposed to preserve the soft and hard tissues in the esthetic zone. These techniques include proper 3D implant positioning, flapless approach, the addition of bone graft, the use of grafts containing growth factors such as concentrated growth factor (CGF) and platelet-rich fibrin (PRF) membranes, the application of connective tissue grafts (CTG), the socket shield technique, or the use of customized healing abutments. In order to offset the peri-implant tissue reduction, various treatments were also devised, including vestibular socket therapy, the dual-zone concept (DZ), and immediate dentoalveolar restoration.

From the above-mentioned approaches, Dual Zone technique was utilized in conjunction with CTG, and CGF graft were primarily advised for peri-implant soft tissue phenotypic preservation, stability, and health. The dual-zone (DZ) concept was developed to reduce the amount of buccal contour change at the extraction site while enhancing the thickness of the peri- implant soft tissues by filling the buccal gap with bone graft in two zones: the bone zone up to the crest of the socket bone and the soft tissue zone. To illustrate, graft particles are absorbed into tissues, increasing their thickness while also providing stability and maintaining soft tissue volume. As a result, the DZ concept aims to maintain the gingival contour while providing excellent soft tissue esthetics.

Connective tissue graft (CTG) and concentrated growth factor (CGF) graft are two commonly used materials for soft tissue augmentation in implant dentistry. CTG has a long history of success in improving soft tissue volume and quality around dental implants by forming a scaffold for cell migration and tissue regeneration. On the other hand, CGF, a newer autologous platelet concentrate rich in growth factors, has demonstrated promising results in stimulating tissue healing and regeneration, potentially outperforming standard graft materials.

To begin with, the success of utilizing CTG in covering exposed roots and increasing the width of the keratinized mucosa (WKM) prompted research into its usage in conjunction with immediate dental implants to improve their final esthetic effects. CTG is thought to be the gold standard for dimensional stability together with IIP in the esthetic zone. Furthermore, inserting CTG concurrently with IIP was claimed to reduce the likelihood of advanced mid-facial mucosal recession, prevent papillae loss, improve soft tissue contour, and reduce crestal bone resorption independent of tissue biotype. Other researches, however, argued that using CTG resulted in bone resorption and lost dimensional stability over time.

Platelets naturally produce Growth factors (GF) such as platelet-derived GF, Transforming GF (TGF)-β1 and β2 (TGF-β2), fibroblast GF, vascular endothelial GF, and insulin-like GF, which promote cell proliferation, matrix remodeling, and angiogenesis. Concentrated GF (CGF) is prepared by centrifuging venous blood, which concentrates platelets in a gel layer made up of a fibrin matrix rich in GFs and leukocytes. CGF operates by degranulating alpha granules in platelets, which play an important role in early wound healing. CGF has been shown to contain more GFs than other platelet-based preparations such as platelet rich fibrin (PRF) and platelet-rich plasma (PRP), and unlike PRP, CGF does not dissolve quickly after application. Furthermore, it was demonstrated that CGF may release GFs for at least 13 days.

CGF, first introduced by Sacco, has recently gained popularity. It is produced by centrifugation of venous blood, similar to PRF, but at a different speed (2400-2700 rpm) to separate cells in the venous blood, resulting in fibrin rich blocks that are much larger, denser, and richer in GF than common PRF. This demonstrates improved regeneration capacity and versatility when utilizing the fibrin-rich block. Furthermore, many studies showed that CGF has higher tensile strength, more growth factors, higher viscosity, and adhesive strength than PRF. As a result, surgeons can utilize CGF as a barrier membrane to speed up soft tissue healing or mix it with bone graft to expedite new bone growth.

Despite the growing interest in immediate dental implants and soft tissue augmentation techniques, limited comparative evidence exists regarding the efficacy of different grafting materials in the dual zone approach, particularly in the esthetic zone. Therefore, there is a need for well-designed randomized controlled clinical trials to evaluate the comparative effectiveness of CTG and CGF grafts in immediate dental implants using the dual zone technique.

This randomized clinical trial aims to address this gap in the literature by comparing the clinical and radiographic outcomes of immediate dental implants with dual zone technique using CTG versus CGF graft in the esthetic zone. By assessing parameters such as volumetric soft tissue alterations, pink esthetic score, clinical measurements, and radiographic bone dimensional changes, this study aims to provide evidence-based guidance for clinicians in selecting the most appropriate grafting material for achieving optimal esthetic outcomes in implant dentistry.

III. Research Question:

Are soft and hard tissue changes following immediate implant placement with dual zone concept and concentrated growth factor graft the same as dual zone concept and connective tissue graft on volumetric analysis, pink esthetic score, clinical, and radiographic measures at baseline, 6 months, and 1 year?

PICOTS Elements:

Patient/Problem :Patients with hopeless teeth requiring extraction in maxillary esthetic zone.

Intervention : Guided immediate implant placement with dual zone technique using concentrated growth factor graft Comparator : Guided immediate implant placement with dual zone technique using connective tissue graft Outcome: Volumetric analysis, Pink Esthetic Score (PES), clinical assessment and radiographic assessment. Time: Baseline and 6 months. Setting : Faculty of Dentistry, Ain Shams University.

ELIGIBILITY:
Inclusion Criteria:

* Systemically (medically) free individuals were recruited for the present study according to the modified Burkett's health history questionnaire, ASA.
* Males and females with age range 20 - 50.
* Patients having a history of hopeless tooth in esthetic zone (Anteriors/Premolars) indicated for extraction and immediate implant placement.
* Patients who are cooperative and maintain proper oral hygiene.
* Intact interproximal and palatal bone extending at least 6 mm apically, with sufficient apical bone to attain implant primary stability (a minimum of 35 Ncm insertion torque).

Exclusion Criteria:

* Heavy smokers. 20
* Patients who exhibit parafunctional occlusal habits 21
* Pregnant ladies or lactating mothers.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Volumetric analysis | Baseline and 6 months
  3D viewer soft tissue; mm changes in the buccal soft tissue contour in comparison to the original ones, at 2,4 and 6 mm from the pre-operative gingival margin

SECONDARY OUTCOMES:
Pink Esthetic Score | 6 months after final crown placement
  This scoring system has seven domains: mesial papilla, distal papilla, soft tissue level, contour, deficient alveolar process, soft tissue color, and texture. Each domain is rated from 0 to 2, with 2 being the highest score. The total PES is the sum of the seven domains' scores, which range from 0 to 14 (14 is the best score, signifying almost identical appearance to the contralateral natural tooth)
Radiographic CBCT measurements | Baseline and 6 months
  Amount of bone labial to implant, horizontal labio-palatal bone reduction, and crestal bone level changes.
Full-mouth plaque score | Baseline and 6 months
  Measured pre-extraction and after 6 months 2 = visible deposit,
  1 = deposit on probing, 0 = no deposit
Full-mouth bleeding score | Baseline and 6 months
  score 0 -normal gingiva; score 1 -mild inflammation, slight change in color, slight oedema, no bleeding on probing; score 2 -moderate inflammation, redness, oedema, and glazing, bleeding on probing; score 3 -severe inflammation, marked redness and oedema, ulceration tendency to spontaneous bleeding.
Visual Analog Scale | 1, 3, and 7 days after the surgery.
  Visual Analog Scale will be recorded by the patient 1, 3, and 7 days after the surgery.
  The patients marked the pain perception in a non-numerical 10 cm line ranging from "no pain = 0" (left) to "very painful = 10" (right).
  1-3 = mild pain 4-6 = moderate pain 7-10 = severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt